CLINICAL TRIAL: NCT01729065
Title: A Randomized Study to Assess the Efficacy of Early Physical Therapy Intervention on Upper Quarter Strength and Mobility, and Reported Upper Extremity Disability and Quality of Life Measures Following a Modified Unilateral Neck Dissection for Treatment of Head and Neck Cancer
Brief Title: A Study to Assess the Efficacy of Early Physical Therapy Intervention Following a Modified Unilateral Neck Dissection for Treatment of Head and Neck Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Melissa M. Eden, Physical Therapist, Orthopedic Clinical Specialist, Primary Investigator, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 09-007403
Record Dates: First submitted 2012-11-09; First posted 2012-11-20 (Estimated); Last update posted 2015-05-22 (Estimated); Status verified 2015-05

CONDITIONS: Shoulder Weakness Following Neck Dissection Surgery
Keywords: Spinal Accessory Nerve Palsy, Cranial Nerve XI, shoulder weakness, neck stiffness, head and neck cancer, neck dissection
MeSH Terms: conditions — Head and Neck Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Home Program (No Intervention): Participants perform home program only.
- Physical Therapy Intervention (Experimental): Physical therapy intervention provided for first 12 weeks following surgery.
  Interventions: Other: Physical therapy intervention

INTERVENTIONS:
Other: Physical therapy intervention — Exercises addressing cervical range of motion, shoulder range of motion and strengthening and scapular stabilization.
  Arms: Physical Therapy Intervention

SUMMARY:
This study will determine whether patients who receive regular physical therapy immediately following a modified neck dissection surgery will report decreased shoulder disability, decreased pain, improved or maintained shoulder range of motion and strength, and improved quality of life than those who receive only home instruction.

ELIGIBILITY:
Inclusion Criteria:

* Adults age 18-85, able to give informed consent
* Subject has provided written informed consent
* Received Modified Unilateral Neck Dissection with sparing of the SAN
* Not currently using transcutaneous electrical nerve stimulation (TENS) as a pain relieving modality
* Not currently receiving acupuncture as a pain relieving modality
* Able to participate with treatment group protocol including physical therapy appointment every other week

Exclusion Criteria:

* History of prior shoulder injury or surgery including rotator cuff repair or total shoulder arthroplasty.
* History of CVA with hemi paresis
* Bilateral neck dissection
* Known severed SAN

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2010-01; Primary Completion 2015-05 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
Disability of the Arm Shoulder and Hand | 12, 24, 36 weeks
  A standardized outcome tool which will be used to measure change in the level of disability related to involvement of the upper extremity at 12, 24, and 36 weeks compared to baseline.

SECONDARY OUTCOMES:
SF-36 | 12, 24, 36 weeks
  General health survey.

OTHER OUTCOMES:
Visual Analog Scale | 12, 24, 36 weeks
  Pain Scale
Strength, range of motion of the neck and shoulder | 12, 24, 36 weeks
  Measurements of shoulder range of motion and strength, cervical range of motion

CONTACTS AND LOCATIONS:
Overall Officials: Melissa M Eden, PT, DPT, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Phoenix, Arizona, United States